CLINICAL TRIAL: NCT02023515
Title: Comparison of Two Programs for Weight Loss and Impact on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kelly Webber (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Kelly Webber, Faculty, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R56HL116517-01A1 (NIH); 1R56HL116517-01A1 (NIH)
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Metabolic Syndrome
Keywords: weight loss; metabolic syndrome; stress; obesity
MeSH Terms: conditions — Metabolic Syndrome; Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress Management (Experimental): Approximately half of the participants will be randomized to a stress management arm. Participants will undergo Emotional Brain Training during a 90 minute session once per week for ten weeks in order to rewire the brain and improve stress management techniques.
  Interventions: Behavioral: Emotional brain training
- standard behavioral weight loss (Active Comparator): Half of participants will receive a standard behavioral weight loss program in 90 minute sessions once per week for 10 weeks
  Interventions: Behavioral: Behavioral weight loss

INTERVENTIONS:
Behavioral: Emotional brain training — Stress management based program
  Arms: Stress Management
Behavioral: Behavioral weight loss — Standard behavioral weight loss
  Arms: standard behavioral weight loss

SUMMARY:
The purpose of this study is to learn the impact stress may have on weight management and emotional eating.

DETAILED DESCRIPTION:
The investigator's long-term goal is to contribute to the development of empirically-based, clinically-useful weight loss and weight maintenance interventions. The objective in this application is to obtain proof of feasibility for a weight loss and maintenance intervention that addresses the underlying issue of stress, as an effective approach to long-term weight loss and maintenance. The central hypothesis for this application is that the weight management intervention utilizing stress management skills will produce weight loss and significant improvements in stress and metabolic syndrome biomarkers at 10 and 20 weeks follow-up. This hypothesis was formulated based upon data showing that stress is associated with increased risk of obesity and a few small studies that have shown this method of stress management can produce long-term weight loss and maintenance and decreased depression and stress. The rationale for the proposed studies is that proof of feasibility for such an intervention will enable subsequent definitive studies at the R01 level. If, however, the investigators were to unexpectedly disprove the concept, such a result would also be valuable because it would lead the investigators to shift focus and redistribute resources accordingly. To test the central hypothesis, and thereby accomplish the objective for this application, the following specific aims will be pursued:

1. Compare a stress management based program to a standard behavioral weight loss program for weight loss and cost-effectiveness. The approach will involve two different intervention groups. Group 1(control) will receive a standard behavioral weight loss program. Group 2 will receive a stress management based intervention built on research in neuroscience and principles of the attachment theory.
2. Determine secondary outcomes from both interventions, including stress as measured by the perceived stress scale. It is hypothesized that Group 2 will show greater improvements in stress at both 10 and 20 weeks follow-up than Group 1.

At the completion of this study, the investigators expect to determine the type of intervention that produces the greatest weight loss in a community sample at 10 and 20 weeks follow-up. The investigators will also have determined what impact the two interventions have on secondary outcomes, including stress as measured by salivary cortisol and telomere length; depression, disordered eating patterns, dietary intake, and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* be 25-55 years of age
* have a BMI of > 28 and <45
* meet criteria for at least one additional risk factor for metabolic syndrome (Participants will be screened for waist circumference and blood pressure to ensure inclusion in the study.)
* own and use a smart phone.

Exclusion Criteria:

* have a medical diagnosis of orthopedic or joint problems that may prohibit regular exercise
* endorse any of the first three items on the Physical Activity Readiness Questionnaire (PAR-Q): heart problems, chest pain, faintness or dizzy spells
* endorse any of the other items on the PAR-Q without a physician's consent
* have had a hospitalization for a psychiatric disorder within the last year
* have a history of anorexia or bulimia nervosa
* have a medical diagnosis of cancer or HIV
* have a diagnosis of a major psychiatric disorder (i.e. bipolar disorder or schizophrenia) or taking anti-psychotic medications
* be pregnant, nursing, or planning to become pregnant within the study period
* be less than 9 months post-partum
* have a weight loss of > 10 pounds in the last six months
* be on more than two medications for hypertension control
* greater than stage 3 kidney disease
* be taking insulin to control diabetes
* be taking Coumadin
* be taking Lasix
* anyone, who in the opinion of the study investigators, would not be a good candidate for the study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly H Webber, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stress Management | Standard Behavioral Weight Loss
Started | 24 | 25
Completed | 23 | 22
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stress Management | Standard Behavioral Weight Loss | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 25 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (8.0) | 44.0 (8.8) | 45.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: Weight change from baseline to 20 weeks
Time Frame: Weight change from baseline to 20 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Stress Management | Standard Behavioral Weight Loss
Number analyzed (Participants) | 24 | 25
kg | 1.6 (3.8) | 3.9 (3.3)

2. Secondary Outcome: Decrease in Stress
Description: Stress was measured by the Perceived Stress Scale (PSS). This scale measures stress on a scale of 0 to 40 points. The results are reported as a total score on the scale. Higher numbers indicate more stress than lower numbers.
Time Frame: PSS change from baseline to 20 weeks
Measure: Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | Stress Management | Standard Behavioral Weight Loss
Number analyzed (Participants) | 24 | 25
units on a scale | -4.5 [-6.8 to -2.2] | -1.8 [-4.5 to 0.9]

ADVERSE EVENTS:
Arm/Group | Stress Management | Standard Behavioral Weight Loss
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No